CLINICAL TRIAL: NCT02313922
Title: Optimizing Psoriasis Treatment of Etanercept Combined Methotrexate: a Phase IV, Multicenter, Randomized, Double-blind, Controlled Trial
Brief Title: Optimizing Psoriasis Treatment of Etanercept Combined Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai CP Guojian Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Min Zheng, director of dermatology, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C301-PS
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- etanercept combined with methotrexate (Experimental): patients treated with etanercept combined with methotrexate
  Interventions: Drug: etanercept combined with methotrexate or etanercept combined with placebo
- etanercept as monotherapy (Experimental): patients treated with etanercept combined with placebo
  Interventions: Drug: etanercept combined with methotrexate or etanercept combined with placebo

INTERVENTIONS:
Drug: etanercept combined with methotrexate or etanercept combined with placebo

SUMMARY:
The purpose of this study is to evaluate whether etanercept combined with methotrexate are superiority than etanercept as monotherapy in the treatment of chinese severe plaque psoriasis. A phase IV, multicenter, randomized, double-blind, controlled trial was conducted.The primary outcome was Change from baseline in plaque psoriasis as assessed by PASI (psoriasis area and severity index) response or PASI75 (a patient that has an improvement from baseline PASI of at least 75%)

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, at least 18 years of age
* have stable plaque psoriasis for at least 6 months, psoriasis involving at least 10 percent of the body surface area, had a minimal PASI of 10 at screening
* had previously received phototherapy or systemic psoriasis therapy at least once or candidates for such therapy in the opinion of the investigator

Exclusion Criteria:

* Patients with guttate, erythrodermic, or pustular psoriasis at the time of screening
* recent infection or opportunistic infections, active tuberculosis, hepatitis B and so on
* liver and kidney dysfunction
* those with other serious, progressive, uncontrolled disorders of vital organs and systems (including cardiovascular, liver, lung and kidney), other autoimmune diseases, cancer, HIV infection, which are not suitable for participation in the study of the disease
* history of significant methotrexate toxicity or total cumulative methotrexate exposure > 1000 mg (unless grade ‡ IIIb liver injury has not occurred)
* use of ultraviolet (UV) B therapy, topical ciclosporin or calcineurin inhibitors, class III through VII topical corticosteroids (permitted on the scalp, axillae, and ⁄or groin), or topical vitamin A or D analogues within 14 days of screening
* and psoralen or UVA therapy, systemic psoriasis therapy (including methotrexate), oral retinoids, class I or II topical corticosteroids, dithranol, cyclophosphamide, sulfasalazine, or intravenous or oral calcineurin inhibitors within 28 days of screening
* Patients were excluded if they had received a tumor necrosis factor (TNF) blocking agent or other biologics within 3 months or interleukin (IL)-12 or IL-23 inhibitors within 6 months of study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2014-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
psoriasis area and severity index 75(PASI75) | 24 weeks
  Change from baseline in plaque psoriasis as assessed by PASI (psoriasis area and severity index) response or PASI75 (a patient that has an improvement from baseline PASI of at least 75%)

SECONDARY OUTCOMES:
psoriasis area and severity index 50(pasi 50) | 24 weeks
  Change from baseline in plaque psoriasis as assessed by PASI (psoriasis area and severity index) response or PASI50 (a patient that has an improvement from baseline PASI of at least 50%)
psoriasis area and severity index 90(pasi 90) | 24 weeks
  Change from baseline in plaque psoriasis as assessed by PASI (psoriasis area and severity index) response or PASI90 (a patient that has an improvement from baseline PASI of at least 90%)
Dermatology Life Quality Index (DLQI) change | 24 weeks
  Change from baseline in plaque psoriasis as assessed by DLQI (dermatology life quality index ) response
adverse events(AEs) | 24 weeks
  Laboratory parameters, rates of AEs, and percentage of patients requiring interruption or discontinuation of study drug due to AEs

CONTACTS AND LOCATIONS:
Locations (1):
- the 2Nd Affiliated Hospital,Zhejiang University,, Hangzhou, Zhejiang, China